CLINICAL TRIAL: NCT02197962
Title: Efficacy of Radial Shockwave Therapy for Treatment of Pain in Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marta Imamura (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor-Investigator, Marta Imamura, Medical Doctor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Radial Shockwave
Record Dates: First submitted 2014-07-17; First posted 2014-07-23 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Radial shockwaves
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extracorporeal radial shockwaves (Experimental): Patients will receive 2,000 impulses of extracorporeal radial shockwave per week, with pressure of 2.5bar to 4.0bar, at the frequency of 8Hz. The impulses will be applied at the most painful site of the knee joint interface on manual palpation, for three consecutive weeks.
  Interventions: Device: Extracorporeal Radial shockwaves
- Placebo Radial Shockwaves (Placebo Comparator): Patients will receive 2,000 impulses of placebo radial shockwave per week, without any energy flow intensity. Frequency of 8Hz will appear in the screen. The impulses will be applied at the most painful site of the knee joint interface on manual palpation, for three consecutive weeks.
  Interventions: Device: Placebo Radial Shockwaves

INTERVENTIONS:
Device: Extracorporeal Radial shockwaves — Patients will receive 2,000 impulses of extracorporeal radial shockwaves or per week, with pressure of 2.5bar to 4.0bar, at the frequency of 8Hz. The impulses will be applied at the most painful site of the knee joint interface on manual palpation, for three consecutive weeks.
  Arms: Extracorporeal radial shockwaves
Device: Placebo Radial Shockwaves — Patients will receive 2,000 impulses of placebo extracorporeal radial shockwaves per week, without any pressure, therefore no energy will be applied, at the frequency of 8Hz. The impulses will be applied at the most painful site of the knee joint interface on manual palpation, for three consecutive weeks.
  Arms: Placebo Radial Shockwaves

SUMMARY:
The objective of this study is to compare the results of 2000 impulses of radius shockwaves per week with 2000 placebo shockwaves on the treatment of pain and functional incapacity of patients with severe primary knee osteoarthritis, who did not satisfactory respond to previous conventional treatments.

DETAILED DESCRIPTION:
* Prospective, placebo controlled randomized and double-blind study.
* Treatment Method:

Radial extracorporeal shockwaves will be applied using the Swiss Dolorclast (EMS Electro Medical Systems, Switzerland), generated by pneumatic waves.

Intervention:

* Group 1 - Intervention group Patients will receive 2,000 impulses of radial shockwave per week, with pressure of 2.5bar to 4.0bar, at the frequency of 8Hz. The impulses will be applied at the most painful site of the knee joint interface on manual palpation, for three consecutive weeks.
* Group 2 - Control Group:

Patients will receive 2,000 impulses of placebo radial shockwave per week, without any energy flow intensity. Frequency of 8Hz will appear in the screen. The impulses will be applied at the most painful site of the knee joint interface on manual palpation, for three consecutive weeks.

Post application program for both groups: Three consecutive days of:

1. Hot packs (superficial heat) applied on the application site for 20 minutes;
2. Simple analgesics, when needed (Acetaminophen 500mg every 6 hours, or analogue in case of allergy).

Outcome Evaluation:

The evaluation of pain intensity will be done according to the VAS (Visual Analog Scale) The influence of pain on the functional capacity of patients will be measured with WOMAC (Western Ontario and McMaster Osteoarthritis Index) for knee evaluation.

Another evaluation criteria will be the level of tolerance of pressure on several muscles and other parts as the pes anserinus and patellar tendon, the knee joint interface, and the supraspinal of L1 to S1 also on the dermatomal from T12 to S2. These measures will be done by the Fisher algometry.

The evaluations will be carried out before the treatment, immediately after the treatment and 3 months after the end of the treatment.

Analgesia drut will be prescribed, if patients feel pain during the days after the application.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of primary knee diagnosis.
* Pain intensity: Visual Analog Scale (VAS) ≥ 6;
* One of more failures with conventional treatment (drugs, Non-Steroidal Anti-inflammatory Drugs - NSAD, physiotherapy, stretching, acupuncture, orthosis and others);
* Age over 60 years;
* No use of corticosteroids in the prior 48 hours;
* No major osteoarthritis events in other joints of lower limbs (waist and ankle) and lower back;
* No clinical evidence of related neuropathy, including radiculopathy and peripheral neuropathy;
* Absence of systemic inflammatory disease (Rheumatoid arthritis, Reiter, ankylosing spondylitis, generalized polyarthritis, cancer);
* Absence of infection or cancer at the application site;
* Absence of related endocrine and metabolic diseases;
* Absence of fibromyalgia, diagnosed after the American College of Rheumatology, 1999;
* Absence of severe blood dyscrasias;
* Absence of severe psychiatric disturbances that requires psychiatric assessment;
* Availability to comply with the clinic visits and follow up evaluations along the treatment

Exclusion Criteria:

* Patients who withdraw the informed consent form at any time

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Before intervention and after 3 months of the end of intervention
  The Visual Analog Scale consists of a straight line of 10cm length which presents the phrase "absence of pain" (0) at one extremity, and unbearable pain (10) at the other extremity.

SECONDARY OUTCOMES:
Level of tolerance of pain | Immediately before the intervention, immediately after the intervention and 3 months after the intervention.
  Measures will be taken with the Fisher algometry in the following muscles: vastus medialis, vastus lateralis, rectus femoris, gracilis, adductor longus, tibialis anterior, fibularis longus, quadratus lumborum, iliopsoas and popliteus; also at the pes anserinus and patellar tendon, the knee joint interface, the supraspinal of L1 to S1 and on the dermatomal from T12 to S2.

OTHER OUTCOMES:
The influence of pain over the functional capacity of patients based on the WOMAC questionnaire | Immediately before the intervention and 3 months after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Imamura, MD, Principal Investigator — Instituto de Medicina Fisica e Reabilitacao HCFMUSP
Locations (2):
- Brazil (2):
  - Instituto de Ortopedia e Traumatologia HCFMUSP, São Paulo, São Paulo
  - Instituto de Medicina Fisica e Reabilitacao HCFMUSP, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No